CLINICAL TRIAL: NCT06170203
Title: Evaluation of the Implementation of Personalised Follow-up in Head and Neck Cancer
Acronym: EMPOWER
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 320336
Record Dates: First submitted 2023-11-28; First posted 2023-12-14 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Personalised Follow-up Pathway — Discharge from routine oncology Follow-Up 2 years following radical treatment for a head and neck cancer

SUMMARY:
The NHS Long Term Plan for Cancer has set out the strategy to deliver personalised care to every patient treated for cancer (1) to improve experience and quality of life for patients. Personalised Follow-Up (PFU) focuses on the tailored needs of patients who have completed cancer treatment and PFU programmes have been established nationally for patients with breast and colorectal cancer. PFU for Head and Neck Cancer (HNC) services will be established nationally by 2024. Currently, there is a lack of evidence that measures prospectively the impact of PFU on patients and providers.

In January 2022, Guys and St. Thomas' NHS Foundation Trust initiated PFU for patients with HNC. For the first 2 years following treatment, patients treated curatively are followed up according to institutional protocol. At 2 years following completion of treatment, patients who remain disease free, have no significant risk factors for recurrence and no severe treatment-related toxicity are referred to the programme and discharged from routine oncology FU. Patients are reviewed in a nurse-led HNC PFU clinic where they receive personalised survivorship, health promotion and education in identifying signs of disease recurrence with information on the pathway to re-present directly to the services at Guy's Cancer.

This mixed methods research project will evaluate implementation factors of this new PFU programme whilst prospectively measuring its effectiveness. A hybrid type 2 implementation-effectiveness study design will be used to determine the value patients and health care providers (HCP). Semi-structured interviews and focus groups with patients and HCP will be undertaken to evaluate barriers and facilitators, safety, acceptability and user experience. Data will be collected over a 24 month period. All patients who are transferred to the PFU pathway will be eligible to participate, alongside HCP involved in delivering the service.

DETAILED DESCRIPTION:
This mixed methods implementation science study aims to develop an understanding of the barriers and facilitators of a high level of fidelity that is sustainable for use by patients and health care providers.

Central to the construct of ethical research is the protection of participants' rights and prevention of harm. Participants should not feel coerced to participate and careful consideration has been given to the recruitment process to ensure informed consent. All participants will be provided with study information at least 10 days before written consent is obtained and verbal consent will be reconfirmed throughout the research process. Participation will be voluntary. Confidentiality of all information will be maintained in accordance with Caldicott Principles. Any patient-identifiable information and research data that is collected will be stored securely on a password-protected encrypted device, in accordance with General Data Protection Regulations. Research data will be collected on paper or electronic web based questionnaires and from qualitative interviews. Primary research data (eg. verbatim transcripts and tabulated data from individual questionnaire responses) will only be accessible to the research team, who are employed by the hospital site.

All patients within the PFU programme will be considered for inclusion within the research, however purposive sampling will be used to select patients for interview to ensure a range of patient demographics, treatments and clinical condition. The researcher will explain the study to patients and will provide a study information pack, including an introductory letter, information sheet and consent form. The researcher will contact the patient at least 48 hours after initial contact to explain the research further and to confirm if the patient would like to participate.

A Patient and Public Involvement (PPI) group comprised of patients and carers' who have received treatment for HNC, has been established to provide expert advice and act in partnership with the researchers with regards to all aspects of the project. PPI members meet bi-monthly to support pathway implementation and will co-design interview schedules to ensure they are participation friendly and ethically sound. PPI members will play a crucial role in ensuring the results of this research are provided with sensitivity to study participants and the wider public once the research is complete.

ELIGIBILITY:
Patient inclusion criteria

* Patients referred to the Head and Neck Cancer Personalised Follow Up clinic
* Patients who had oncological treatment for a Head and Neck cancer
* Patients who were treated with curative intent and who are disease free
* Patients who are at least 2 years post treatment completion
* Patients who have no risk factors of disease recurrence Staff Criteria
* Oncologists, surgeons, allied health practitioners, nurses, and support staff who provide care for patients with Head and Neck Cancer
* Willing to participate in a qualitative interview or focus group

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who have been treated for Head and Neck Cancer. Members of the MDT caring for patients who have been treated for HNC
Sampling Method: Non-Probability Sample
Enrollment: 33 (Estimated)
Dates: Start 2023-08-08 (Actual); Primary Completion 2024-09-10 (Estimated); Study Completion 2024-09-10 (Estimated)

PRIMARY OUTCOMES:
Acceptability of PFU pathway to patients with Head and Neck Cancer. | End of study, 12 months
  Semi structured interviews will be conducted with patients within the Personalised Follow Up Pathway to explore the acceptability of the pathway, the resources and the transition of care away from the 5 year follow up pathway
Acceptability of PFU pathway to service providers within Head and Neck Cancer. | End of study, 12 months
  Semi structured interviews will be conducted with service providers within Head and Neck Cancer, to explore the acceptability of the pathway, the resources and the protocol.
Safety of a Personalised Follow Up Pathway within Head and Neck Cancer | End of study, 12 months
  Clinical data will be collected with regards to any recurrent cancers that are diagnosed for patients within this pathway. Time from symptom recognition to clinical review and diagnosis will be monitored.

SECONDARY OUTCOMES:
Patient experience within the Personalised Follow Up Pathway. | End of study, 12 months
  Cross sectional patient surveys and semi-structured interviews will be conducted to explore the experience of patients within the Personalised Follow Up Pathway
Service provider experience within the Personalised Follow Up Pathway. | End of study, 12 months
  Semi-structured interviews will be conducted to explore the experience of service providers within the Personalised Follow Up Pathway.
Sustainability of the Personalised Follow Up Pathway | End of study, 12 months
  Semi structured interviews will be conducted with patients and staff to explore the barriers and facilitators that will influence the sustainability of this pathway, within the institution

CONTACTS AND LOCATIONS:
Locations (1):
- Laura Dean, London, United Kingdom

REFERENCES:
- [Background] 1. NHS England. The NHS Long Term Plan. (2019) https://www.longtermplan.nhs.uk